CLINICAL TRIAL: NCT00001812
Title: A Randomized, Double-Blind, Placebo Controlled Trial Evaluating the Impact of Nystatin on the Development of Oral Irritation in Patients Receiving High Dose Intravenous Interleukin-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990097; 99-C-0097
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Candidiasis, Oral; Gastrointestinal Diseases; Stomatitis
Keywords: Mucositis; Oral Candidiasis; Prophylaxis; Stomatitis; Swish and Swallow
MeSH Terms: conditions — Candidiasis, Oral; Gastrointestinal Diseases; Stomatitis; Mucositis | interventions — Nystatin

INTERVENTIONS:
Drug: Nystatin

SUMMARY:
In patients who are receiving intravenous high dose Interleukin-2, patients will be randomized into two groups: group one will receive nystatin swish and swallow immediately before initiation of IL-2, and the second group will receive a placebo. The patients in each group will be monitored and evaluated for differences in the rate and severity of development of oral irritation during treatment. They will also be studied for differences between the two groups in the number of doses of IL-2 taken.

DETAILED DESCRIPTION:
In patients who are receiving intravenous high dose Interleukin-2, patients will be randomized into two groups: group one will receive nystatin swish and swallow immediately before initiation of IL-2, and the second group will receive a placebo. The patients in each group will be monitored and evaluated for differences in the rate and severity of development of oral irritation during treatment. They will also be studied for differences between the two groups in the number of doses of IL-2 taken.

ELIGIBILITY:
All patients enrolled on high dose intravenous interleukin-2 studies in the Surgery Branch of the National Cancer Institute are eligible, except for patients who are receiving adoptively transferred cells (cloned peripheral blood cells).

All inclusion criteria as stated in the parent immunotherapy protocol apply:

No patients with evidence of oral irritation prior to starting therapy;

No patients with any known sensitivity to nystatin;

No patients receiving systemic antifungals;

No patients with active oral infections.

In additional, all exclusion criteria as stated in the parent immunotherapy protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84
Dates: Start 1999-04; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Marmary Y, Shiloni E, Katz J. Oral changes in interleukin-2 treated patients: a preliminary report. J Oral Pathol Med. 1992 May;21(5):230-1. doi: 10.1111/j.1600-0714.1992.tb00107.x. PMID 1403839
- [Background] Rodriguez-Archilla A, Urquia M, Cutando A, Asencio R. Denture stomatitis: quantification of interleukin-2 production by mononuclear blood cells cultured with Candida albicans. J Prosthet Dent. 1996 Apr;75(4):426-31. doi: 10.1016/s0022-3913(96)90036-0. PMID 8642530
- [Background] Rosenberg SA, Lotze MT, Muul LM, Leitman S, Chang AE, Ettinghausen SE, Matory YL, Skibber JM, Shiloni E, Vetto JT, et al. Observations on the systemic administration of autologous lymphokine-activated killer cells and recombinant interleukin-2 to patients with metastatic cancer. N Engl J Med. 1985 Dec 5;313(23):1485-92. doi: 10.1056/NEJM198512053132327. PMID 3903508